CLINICAL TRIAL: NCT06310447
Title: Determination of Ecological Awareness and Attitudes Levels of Undergraduate Students Studying in The Physiotherapy and Rehabilitation Department in Istanbul
Brief Title: Determination of Ecological Awareness and Attitudes Levels of Undergraduate Physiotherapy Students in Istanbul
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Elif Elcin Dereli, Principal Investigator, Istanbul Bilgi University
Other Study IDs: IstanbulBUFC2
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Ecological and Environmental Concepts
Keywords: ecological awareness; ecological attitude; physiotherapy and rehabilitation; carbon footprint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students: Students of the physiotherapy and rehabilitation department in Istanbul constitute the population of the research.

SUMMARY:
The natural environment, which is the living environment of all living things; Technological advances and industrialization activities are being affected more and more negatively every day. Increasing energy demand and resource consumption due to population growth lead to negative consequences on ecological balance, such as environmental pollution, climate change and loss of natural environments. Health services have also increased resource use with the advancement of technology and caused negative effects on the environment. Health services have been slow to understand their impact on the environment. The aim of the study is to determine the environmental awareness and environmental attitude levels of physiotherapy and rehabilitation department students, to popularize the field of "Environmental Physiotherapy" and to enable the training of physiotherapist candidates with high environmental awareness.

DETAILED DESCRIPTION:
The natural environment, which is the living environment of all living things; Technological advances and industrialization activities are being affected more and more negatively every day. Increasing energy demand and resource consumption due to population growth leads to negative consequences on ecological balance, such as environmental pollution, climate change and loss of natural environments. Health services have also increased resource use with the advancement of technology and caused negative effects on the environment. Health services have been slow to understand their impact on the environment. The aim of the study is to determine the environmental awareness and environmental attitude levels of physiotherapy and rehabilitation department students, to popularize the field of "Environmental Physiotherapy" and to enable the training of physiotherapist candidates with high environmental awareness. In this descriptive study planned on physiotherapy and rehabilitation department students studying in Istanbul, participants who meet the inclusion criteria and volunteer for the study will be included. "Socio-demographic information form", "Ecological Footprint Awareness Scale", "Environmental Awareness Scale", "Environmental Attitude Scale" and 5-question survey forms prepared by the researchers will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Istanbul
* Being a physiotherapy and rehabilitation undergraduate student
* Being a 2nd, 3rd or 4th grade student
* Volunteering to participate in the study

Exclusion Criteria:

* Being a first year student of physiotherapy and rehabilitation
* Refusing to participate in the study

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: The population of the research consists of 2nd, 3rd and 4th grade undergraduate students studying and living in the physiotherapy and rehabilitation department in Istanbul.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Ecological Footprint Awareness Scale | Baseline
  The scale consists of 30 questions and six subgroups. The subgroups are Energy (questions 1-8), Within the Scope of Laws (questions 9-12), Recycling (questions 13-17), Transportation (questions 18-22), It consists of the headings Food (questions 23-26) and Water Consumption (questions 27-30). Scoring of the scale is obtained by scoring the answers to the survey questions in the range of 1-5 points between Strongly Disagree and Strongly Agree. A validity and reliability study was conducted for the use of the scale. Permission was received via e-mail from the responsible researcher in this validity and reliability study to use the ecological footprint awareness scale in our study.The scale is scored between 30-150. A higher score means higher ecological footprint awareness.
Environmental Awareness Scale | Baseline
  The scale consists of 18 questions. The scoring of the scale, which was created to provide information about the environmental awareness of the people who answered the survey, is achieved by scoring the answers to the survey questions in the range of 1-5 points between "Strongly Disagree" and "Strongly Agree". Permission was received via e-mail from the responsible researcher in the Turkish validity and reliability study to use the environmental attitude scale in our study. The scale is scored between 18-90. A higher score means higher environmental awareness.
Environmental Attitude Scale | Baseline
  The scale consists of 22 questions. The survey was created to obtain information about the environmental attitudes of the people who answered the survey. Scoring of the scale is achieved by scoring the answers to the survey questions in the range of 1-5 points between "Strongly Disagree" and "Strongly Agree". Questions 6, 7, 9, 10, 17, 18, 19, 21 and 22 of the survey questions have reverse coding. Permission was received via e-mail from the responsible researcher in the validity and reliability study to use the environmental attitude scale in our study. The scale is scored between 22-110. A higher score means better environmental attitude.

SECONDARY OUTCOMES:
Participant Information Form | Baseline
  The survey created by the researchers consists of 5 questions. It was prepared to examine whether the participants have knowledge about the field of environmental physiotherapy. (Generally yes/no questions for descriptive data, no scoring.) It questions whether the participant has heard of the concept of environmental physiotherapy, whether the participant has taken courses or read in this field, and their thoughts on this subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided